CLINICAL TRIAL: NCT00862407
Title: Impact of Pulsatile CPB on Vital Organ Recovery
Brief Title: Impact of Pulsatile Cardio-Pulmonary Bypass (CPB) on Vital Organ Recovery
Status: Active, not recruiting | Type: Observational
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: Penn State University (Other)
Responsible Party: Principal Investigator, Akif Undar, Professor of Pediatrics, Surgery, & Bioengineering, Milton S. Hershey Medical Center
Other Study IDs: 19299
Record Dates: First submitted 2009-03-13; First posted 2009-03-16 (Estimated); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Cardio-Pulmonary Bypass
Keywords: Cardiopulmonary bypass; Non-pulsatile perfusion; Pulsatile perfusion; plasma proteins

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Blood and plasma samples
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: Non-pulsatile Group (conventional)
- 2: Pulsatile group (Alternate)

SUMMARY:
This research study is about the effect heart-lung bypass procedures have on the vital organs (brain, heart, lungs, and kidneys) during open-heart surgery in pediatric patients. There are two types of heart pumps used in surgery requiring heart-lung bypass; one pumps the blood continuously through the body and the other pumps the blood with repeated pulses. Both pumps are approved for clinical use by the FDA. Although 90% of institutions still use non-pulsatile flow, some studies show there may be benefits to using pulsatile flow during surgery.

The investigators want to learn whether the vital organs (brain, heart, lungs, and kidneys) respond differently to one method than they do to the other. Approximately 300 children will take part in this research at the Hershey Medical Center.

ELIGIBILITY:
Inclusion Criteria:

* Patients recruited from Penn State Children's Hospital undergoing cardiac surgery with cardiopulmonary bypass.

Exclusion Criteria:

* Patients older than 17 years will be excluded.

Ages: 1 Day to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: 300 children (150 per perfusion system) ages 1 year to < 18 years requiring CPB for cardiac surgery.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2008-10; Primary Completion 2025-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in plasma proteins | 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Penn State College of Medicine, Hershey, Pennsylvania, United States

REFERENCES:
- See also: Pediatric Cardiac Research Laboratories — http://www.pennstatehershey.org/web/childrensheartgroup/research/overview
- See also: International Conference on pediatric heart pumps — http://www.hmc.psu.edu/childrens/pedscpb/